CLINICAL TRIAL: NCT00912652
Title: Rural Lifestyle Intervention Treatment Effectiveness Trial
Acronym: RuralLITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RuralLITE-N; R18HL087800 (NIH)
Record Dates: First submitted 2009-05-29; First posted 2009-06-03 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: obesity; rural health; exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Intensity Lifestyle Intervention (Experimental): High intensity group will receive 48 sessions of lifestyle intervention over a two-year period
  Interventions: Behavioral: lifestyle intervention
- Mod. Intensity Lifestyle Intervention (Experimental): Moderate intensity group will receive 32 sessions of lifestyle intervention over a two-year period.
  Interventions: Behavioral: lifestyle intervention
- Low Intensity Lifestyle Intervention (Experimental): Low intensity group will receive 16 sessions of lifestyle intervention over a two-year period.
  Interventions: Behavioral: lifestyle intervention
- Health Education Control (Active Comparator): Health education control group will receive 16 sessions of health education related to diet and exercise over a two-year period.
  Interventions: Behavioral: Health Education Control

INTERVENTIONS:
Behavioral: lifestyle intervention — Three doses of lifestyle intervention will be compared to an education control condition.
  Arms: High Intensity Lifestyle Intervention; Low Intensity Lifestyle Intervention; Mod. Intensity Lifestyle Intervention
Behavioral: Health Education Control — Health education control group will receive 16 session of health education related to diet and exercise over a two-year period.
  Arms: Health Education Control

SUMMARY:
More and more Americans are becoming overweight. The rates of overweight are especially high in rural areas of the country. Until now, there has been little access to weight management programs in rural areas. This study will examine ways to help individuals from rural counties to manage weight and improve fitness. To do this, three doses of lifestyle treatment (Low, Moderate and High)will be compared to an education control condition. Our principal hypothesis is that both the Moderate and High conditions will have greater weight loss at two years than either the Low or Control conditions.

DETAILED DESCRIPTION:
Higher rates of obesity, sedentary lifestyle, and coronary heart disease are observed in rural than in non-rural areas of the U.S., yet the treatment of obesity in the rural population has received little attention. Efficacy trials, conducted in academic health centers, show that lifestyle interventions can produce sufficient weight reductions to improve health, but very few trials have been carried out in medically underserved community settings. Moreover, the high intensity of treatments used in efficacy studies represents a barrier to dissemination into rural settings. The existing infrastructure of the United States Department of Agriculture Cooperative Extension Service, with over 2900 offices nationwide, may serve as a valuable resource for bringing lifestyle interventions to rural areas. Preliminary data from our rural obesity research program show promising findings for lifestyle interventions delivered through Extension offices. The next logical step in this line of research is to determine the minimum intensity of treatment required to produce clinically meaningful, long-term weight reductions. We propose to conduct a single-blind, multi-site, randomized controlled trial in obese adults (N=542) to evaluate the effects of LOW, MODERATE, and HIGH doses of lifestyle treatment on two-year changes in body weight, compared to an education CONTROL condition. The LOW intensity condition reflects the dose of group treatment commonly used in community settings, whereas the HIGH dose corresponds to the intensity level employed in efficacy trials. The MODERATE intensity intervention represents a treatment dose that our preliminary data suggest may provide benefits comparable to the HIGH intensity intervention. Our principal hypothesis is that both the MODERATE and HIGH interventions will produce greater weight reductions at two years than either the LOW or CONTROL conditions. We will also evaluate the proportion of participants in each condition, who achieve clinically significant weight losses, and we will examine changes in metabolic risk factors, dietary intake, physical activity, and quality of life. We will calculate the cost-effectiveness of the interventions, and we will investigate potential mediators of long-term change.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21 to 75 years
* Body Mass Index: 30 to 45 kg/m**2

Exclusion Criteria:

* Underlying disease likely to limit lifespan and/or increase risk of interventions:cancer requiring treatment in past five years (exception: non-melanoma skin cancer); serious infectious diseases (e.g., self-reported HIV, self-reported tuberculosis or treatment); myocardial infarction or cerebrovascular accident within the last six months; unstable angina within the past six months; congestive heart failure; chronic hepatitis; cirrhosis; chronic malabsorption syndrome; chronic pancreatitis; irritable bowel syndrome; previous bariatric surgery; history of organ transplantation; history of musculoskeletal conditions that limit walking; chronic lung diseases that limit physical activity; and any other condition likely to limit five-year life expectancy.
* Metabolic exclusions: fasting blood glucose > 125 mg/dl at screening if not known to be diabetic (diabetic patients under active treatment will be enrolled if approved by primary provider); fasting serum triglycerides > 400 mg/dl at screening; resting blood pressure > 140/90 mm Hg.
* Medication exclusions: antipsychotic agents; monoamine oxidase inhibitors; systemic corticosteroids; antibiotics for HIV or Tuberculosis; chemotherapeutic drugs; or use of prescription weight-loss drugs within six months.
* Conditions or behaviors likely to affect the conduct of the trial: unwilling or unable to give informed consent; unable to read English at the 5th grade level; unwilling to accept random assignment; unwilling to travel to Extension office for intervention sessions; participation in another randomized research project; weight loss > 10 pounds in past six months; likely to move out of the county in next two years; major psychiatric disorder; excessive alcohol intake; BMI > 45; prior participation in the TOURS trial; and other conditions which in the opinion of staff would adversely affect participation in the trial

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2008-06; Primary Completion 2013-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
body weight | two years

SECONDARY OUTCOMES:
blood pressure | two years
lipid profile | two years
glycemic control | two years
High-sensitivity C-reactive protein (hsCRP) | two years
physical activity | two-years
physical performance | two-years
dietary intake | two-years
waist circumference | two-years
health-related quality of life | two-years

CONTACTS AND LOCATIONS:
Overall Officials: Michael G. Perri, Ph.D., Principal Investigator — University of Florida
Locations (8):
- United States (8):
  - Levy County, Bronson, Florida
  - Flagler County, Bunnell, Florida
  - Dixie County, Cross City, Florida
  - Putnam County, East Palatka, Florida
  - Suwannee County, Live Oak, Florida
  - Baker County, Macclenny, Florida
  - Lafayette County, Mayo, Florida
  - Bradford County, Starke, Florida

REFERENCES:
- [Background] Perri MG, Limacher MC, von Castel-Roberts K, Daniels MJ, Durning PE, Janicke DM, Bobroff LB, Radcliff TA, Milsom VA, Kim C, Martin AD. Comparative effectiveness of three doses of weight-loss counseling: two-year findings from the rural LITE trial. Obesity (Silver Spring). 2014 Nov;22(11):2293-300. doi: 10.1002/oby.20832. PMID 25376396
- [Derived] Radcliff TA, Cote MJ, Whittington MD, Daniels MJ, Bobroff LB, Janicke DM, Perri MG. Cost-Effectiveness of Three Doses of a Behavioral Intervention to Prevent or Delay Type 2 Diabetes in Rural Areas. J Acad Nutr Diet. 2020 Jul;120(7):1163-1171. doi: 10.1016/j.jand.2019.10.025. Epub 2019 Dec 30. PMID 31899170
- [Derived] Bauman V, Ariel-Donges AH, Gordon EL, Daniels MJ, Xu D, Ross KM, Limacher MC, Perri MG. Effect of dose of behavioral weight loss treatment on glycemic control in adults with prediabetes. BMJ Open Diabetes Res Care. 2019 May 28;7(1):e000653. doi: 10.1136/bmjdrc-2019-000653. eCollection 2019. PMID 31245006